CLINICAL TRIAL: NCT03980496
Title: Effects of Different Omeprazole Dosing on Gastric pH in Non- Variceal Upper Gastrointestinal Bleeding: A Randomized Prospective Study
Brief Title: Effects of Different Omeprazole Dosing on Gastric pH in Non-variceal Upper Gastrointestinal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N N402 462539; 4625/B/P01/2010/39 (Other: Polish National Science Centre)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Non-variceal Upper Gastrointestinal Bleeding
Keywords: CYP2C19; Helicobacter pylori; non-variceal upper gastrointestinal bleeding; intragastric pH; proton pump inhibitor
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- omeprazole infusion (OI) group (Active Comparator): After successful endoscopic hemostasis, the patients are given an 80-mg i.v. omeprazole bolus. The OI group is then treated with an 8-mg/h continuous i.v. infusion of OME for 72 h.
  Interventions: Drug: Omeprazole
- omeprazole bolus (OB) group (Active Comparator): After successful endoscopic hemostasis, the patients are given an 80-mg i.v. omeprazole bolus. The OB group receives a 40-mg i.v. bolus of OME every 12 h.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole
  Other Names: endoscopic treatment of non-variceal upper gastrointestinal bleeding

SUMMARY:
The aim of the study is to identify the best method of omeprazole (OME) application with respect to intragastric pH, cytochrome P450 2C19 (CYP2C19) genotype and phenotype.

DETAILED DESCRIPTION:
The patients with non-variceal upper gastrointestinal bleeding (NVUGIB) are prospectively enrolled. After the achievement of endoscopic hemostasis, the patients are randomized to 40-mg intravenous (i.v.) OME bolus injection every 12 h or 8-mg/h continuous i.v. infusion for 72 h after an 80-mg i.v. OME bolus administration. The intragastric pH is recorded for 72 h. The CYP2C19 variant alleles (*2, *3, *17) are analyzed and the serum concentrations of OME and 5-hydroxyomeprazole (5-OH OME) are determined. The diagnosis of Helicobacter pylori infection was based on the results of the rapid urease test performed on stomach mucosa biopsies (antrum and angle) and on the results of the stool antigen test.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent must be obtained before any treatment or assessment is performed
* patients admitted with upper gastrointestinal bleeding (UGIB) symptoms to the Emergency Department of the University Hospital of Bialystok (Bialystok, Poland)

Exclusion Criteria:

* pregnancy
* age >90 years
* lack of written consent
* recent treatment with certain medications, including PPIs, H2-receptor antagonists (H2RA), antacids, steroids, oral contraceptives, clopidogrel, prasugrel and clarithromycin
* the presence of variceal UGIB
* history of surgery of upper gastro-intestinal tract

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09-09 (Actual); Primary Completion 2013-06-08 (Actual); Study Completion 2013-06-08 (Actual)

PRIMARY OUTCOMES:
Intragastric pH in non-variceal upper gastrointestinal bleeding patients treated with omeprazole regarding: Percentage of time at pH >4.0 and pH >6.0 | 72 hours
  intragastric pH profiles
Intragastric pH in non-variceal upper gastrointestinal bleeding patients treated with omeprazole regarding: pH at specified time after the initial OME 80 mg i.v. bolus | 72 hours
  intragastric pH profiles
Intragastric pH in non-variceal upper gastrointestinal bleeding patients treated with omeprazole regarding: Helicobacter pylori infection | 72 hours
  intragastric pH profiles
Intragastric pH in non-variceal upper gastrointestinal bleeding patients treated with omeprazole regarding: CYP2C19 variant alleles (*2, *3, *17) | 72 hours
  intragastric pH profiles

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Dabrowski, Prof., Study Chair — Medical University of Bialystok
Locations (1):
- Department of Gastroenterology and Internal Medicine, Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

REFERENCES:
- [Result] Chwiesko A, Charkiewicz R, Niklinski J, Luczaj W, Skrzydlewska E, Milewski R, Baniukiewicz A, Wroblewski E, Rosolowski M, Dabrowski A. Effects of different omeprazole dosing on gastric pH in non-variceal upper gastrointestinal bleeding: A randomized prospective study. J Dig Dis. 2016 Sep;17(9):588-599. doi: 10.1111/1751-2980.12393. PMID 27518195